CLINICAL TRIAL: NCT01710436
Title: Relationship Between Dosage of Clopidogrel and Platelet Aggregation in Chinese With Different Genotype
Acronym: RDPAC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Xiaoxing Zhang, MD, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: RDPAC2012
Record Dates: First submitted 2012-10-15; First posted 2012-10-19 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-05

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Low dose - Wild genotype (LW): 75mg Qd > 7d Clopidogrel pre-treatment before PCI, according to the reality; CYP2C19 wild genotype
- Low dose - Variant genotype (LV): 75mg Qd > 7d Clopidogrel pre-treatment before PCI, according to the reality; CYP2C19 variant genotype
- High dose - Wild genotype (HW): 300mg Clopidogrel loading dose pre-treatment before PCI, according to the reality; CYP2C19 wild genotype
- High dose - Variant genotype (HV): 300mg Clopidogrel loading dose pre-treatment before PCI, according to the reality; CYP2C19 variant genotype

SUMMARY:
This study is a prospective, observational study to estimate the relationship between dosage of clopidogrel and platelet aggregation in Chinese with different genotype. The investigators suppose both pretreatment dosage of clopidogrel before percutaneous coronary intervention (PCI) and CYP2C19 genotype may effect the platelet aggregation as well as clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* accept PCI in Chinese CHD patients
* expected dual antiplatelet therapy (DAPT) at least 6 months

Exclusion Criteria:

* another planned PCI within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese coronary heart disease (CHD) patient
Sampling Method: Probability Sample
Enrollment: 880 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in platelet aggregation | 1 month and 6 months after PCI

SECONDARY OUTCOMES:
Major adverse cardiovascular events (MACE); Bleeding events | 6 months after PCI

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Institute and Fu Wai Hospital, CAMS & PUMC, Beijing, China

REFERENCES:
- [Derived] Zhang X, Yan L, Wang D, Li Y, Han L, Tian L, Liu H, Li Y. Comparison of loading with maintenance dose of clopidogrel on platelet reactivity in Chinese with different CYP2C19 genotypes prior to percutaneous coronary intervention. Chin Med J (Engl). 2014;127(14):2571-7. PMID 25043069